CLINICAL TRIAL: NCT04353934
Title: The Ariel University Survey on Dietary Changes and Anxiety During the Coronavirus Pandemic: TARUS
Brief Title: The Ariel University Survey on Dietary Changes and Anxiety During the Coronavirus Pandemic
Acronym: TARUS
Status: Completed | Type: Observational
Sponsor: Ariel University (Other)
Responsible Party: Sponsor
Other Study IDs: AU-HEA-VKS-20200329
Record Dates: First submitted 2020-04-12; First posted 2020-04-21 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Dietary Habits; Anxiety
Keywords: Coronavirus pandemic
MeSH Terms: conditions — Feeding Behavior; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Respondents: All adults aged 18 or older who elect to respond to the online survey

SUMMARY:
Background/Objectives: Psychological anxiety has been associated with alterations in eating patterns. The 2020 global coronavirus pandemic has created a situation characterized by increased anxiety. The present international survey was designed to examine associations between exposure to quarantine/isolation measures, anxiety levels and changes in dietary patterns.

Methods: The present study utilizes a Google Survey platform to conduct an international survey querrying dietary patterns before vs. after the coronavirus pandemic; anxiety during the pandemic; and demographic characteristics. The nutrition portion of the survey is based on the Mediterranean Diet Score while the anxiety estimate is based on the GAD-7. The survey is available in English, Hebrew, Spanish, Italian, French, Arabic and Russian. It has been distributed via social media.

Anticipated Results: We believe that changes in dietary habits will be identified and that these will be associated with anxiety levels. Additionally, we believe that by-country differences will be identified.

Discussion: The Google Survey format distributed by social media provides an almost immediate means of distributing the survey globally. The survey can only be completed if the respondent first indicates his/her informed consent. The convenience sample limits generalizability to individuals who volunteer to complete online surveys; however, we anticipate a large response which may mitigate this limitation.

DETAILED DESCRIPTION:
The study will leverage the COVID-19 pandemic to study associations between dietary patterns, weight changes and anxiety.

The study utilizes an online survey, publicized on public and personal social media pages, to query demographics, dietary and exercise patterns and measures of anxiety. Dietary patterns are assessed using the Mediterranean Diet Score, which evaluates the similarity between reported dietary intake and the Mediterranen Diet Pattern, which has been shown to reduce all-cause mortality and cardiovascular morbidity and mortality. Changes in dietary patterns and duration of exercise during vs. prior to the pandemic are measured. Anxiety is measured using the General Anxiety Disorder (GAD)-7 scale. Additional measures of social isolation, both prior to and during the pandemic, are queried in the survey. Data are anonymous and investigators have no ability to associated the response to an individual or IP address. However, interested respondents can provide an email address to which an analysis of the diet score can be sent. Data are automatically downloaded to an Excel spreadsheet, and this is cleaned and uploaded to SPSS for analysis. Continuous data are assessed for normality using the Kolmogorov-Smirnov test and will be summarized using median (IQ range) or mean (sd) as appropriate. Nominal data will be summarized in frequency tables and presented as n (%). Associations between the total Mediterranean Diet Score and the GAD-7 will be described by calculating the Pearson's or Spearman's correlation coefficient as appropriate. Before vs. after responses will be evaluated using the Wilcoxon Signed Ranks Test or the McNemar Test. Differences in responses by demographic characteristics will be measured using the t-test for independent samples, the Mann-Whitney U or ANOVA as appropriate. The GAD-7 score will be dichotomized to moderate anxiety or more (GAD-7=10) vs. lower, and modeled using logistic regression analyisis.

The survey format permits real time response to the ongoing pandemic and the multi-lingual presentation allows for a wide potential population of respondents who can reply in a language in which they are comfortable. Further, this permits by-language comparisons.

ELIGIBILITY:
Inclusion Criteria: All adult individuals (aged 18 or older) who see and elect to respond to the survey will be included.

-

Exclusion Criteria: Subjects who indicate that their age is younger than 18 years, and those who do not provide informed consent will be excluded.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include all adult individuals who see and elect to complete the survey online and who provide informed consent by clicking on the appropriate button.
Sampling Method: Non-Probability Sample
Enrollment: 3797 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
The association between Mediterranean Diet Score and Anxiety Score | through study completion, average six months
  The Mediterranean Diet Score (MedDiet Score) will be calculated and correlated to the Anxiety Score (GAD-7)
The degree to which current dietary intake is consisten with the Mediterranean Diet | through study completion, average six months
  Mediterranean Diet Score (MedDiet) will be calculated

SECONDARY OUTCOMES:
By-country comparisons of the association between Mediterranean Diet (MedDiet) score and Anxiety | through study completion, average six months
  By-country comparisons of the association between Mediterranean Diet (MedDiet) score and Anxiety (GAD-7)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Boaz, RD, PhD, Principal Investigator — Department of Nutrition Sciences, Ariel University
Locations (1):
- Ariel University, Ariel, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abu-Saad K, Endevelt R, Goldsmith R, Shimony T, Nitsan L, Shahar DR, Keinan-Boker L, Ziv A, Kalter-Leibovici O. Adaptation and predictive utility of a Mediterranean diet screener score. Clin Nutr. 2019 Dec;38(6):2928-2935. doi: 10.1016/j.clnu.2018.12.034. Epub 2019 Jan 5. PMID 30642736
- [Background] Esser P, Hartung TJ, Friedrich M, Johansen C, Wittchen HU, Faller H, Koch U, Harter M, Keller M, Schulz H, Wegscheider K, Weis J, Mehnert A. The Generalized Anxiety Disorder Screener (GAD-7) and the anxiety module of the Hospital and Depression Scale (HADS-A) as screening tools for generalized anxiety disorder among cancer patients. Psychooncology. 2018 Jun;27(6):1509-1516. doi: 10.1002/pon.4681. Epub 2018 Mar 30. PMID 29473255
- [Derived] Kaufman-Shriqui V, Navarro DA, Raz O, Boaz M. Multinational dietary changes and anxiety during the coronavirus pandemic-findings from Israel. Isr J Health Policy Res. 2021 Mar 23;10(1):28. doi: 10.1186/s13584-021-00461-1. PMID 33757598
- See also: Survey page — http://da3761.wixsite.com/research